CLINICAL TRIAL: NCT01222195
Title: Phase II Study of Lenalidomide and Darbepoetin Alfa in Myelodysplastic Syndrome (Low to Intermediate-1 Risk Category Excluding 5q Deletion)
Brief Title: Lenalidomide and Darbepoetin in Low-Intermediate Risk Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0657
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia
Keywords: Myelodysplastic Syndrome; Red cell transfusion independence; Darbepoetin alfa; Lenalidomide; CC-5013; Revlimid; Aranesp; Erythropoietin; Erythropoiesis Stimulating Protein
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Lenalidomide; Darbepoetin alfa; Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide + Darbepoetin alfa (Experimental): Lenalidomide 10 mg/day orally days 1-21 and Darbepoetin alfa 200 mcg subcutaneously every 2 weeks of 28 day cycle
  Interventions: Drug: Lenalidomide; Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Lenalidomide — 10 mg/day by mouth on days 1-21 of every 28 day cycle.
  Other Names: CC-5013; Revlimid
Drug: Darbepoetin alfa — 200 mcg subcutaneously every 2 weeks of a 28 cycle.
  Other Names: Aranesp; Erythropoietin; Erythropoiesis Stimulating Protein

SUMMARY:
The goal of this clinical research study is to learn if lenalidomide and darbepoetin alfa given together will help to control the need for transfusions in patients with low to intermediate risk Myelodysplastic Syndrome (MDS). The safety of this combination will also be studied.

DETAILED DESCRIPTION:
Lenalidomide is designed to change the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells. Darbepoetin alfa is designed to stimulate production of red blood cells.

If you are found to be eligible to take part in this study, you will take lenalidomide once a day by mouth on Days 1-21. On Days 22-28, you will not take lenalidomide. Swallow lenalidomide capsules whole with water at the same time each day. Do not break, chew or open the capsules.

If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose).

Due to the uncertain amount of re-absorption of lenalidomide, there will be no re-dose for lenalidomide if you vomit the pills.

Every 28 days is called a study "cycle". Since lenalidomide may cause blood clots, you will take aspirin every day, by mouth, unless your platelet count is too low. Darbepoetin alfa will be given through a needle under the skin (subcutaneously) once every 2 weeks.

You will be given a drug diary. In this diary, you will record when you take the study drugs and any side effects you may have.

During Cycle 1, you will have a study visit just before receiving lenalidomide and then once a month for the first 3 months, then every 3 months after that. At these visits, you will have a physical exam. Blood (about 2 tablespoons) will be drawn for routine tests. Your drug diary will be checked and you will return the bottle of the study drug and any unused drug. You will receive one cycle supply of lenalidomide.

At the end of the first 3 cycles, or earlier if your doctor thinks it is necessary, you will have a bone marrow aspirate. If your doctor thinks it is necessary, you may have additional bone marrow aspirates while on study.

You may remain on study for as long as you are benefitting. You will be taken off study if the disease gets worse or intolerable side effects occur.

Once you are off-study, you will have an end-of-study visit. At this visit, blood (about 2 tablespoons) will be drawn for routine tests. If you are a woman who is able to have children, a portion of this blood will be used for a blood pregnancy test.

You will be contacted by phone 30 days after you are taken off study, and then every 3 months. You will be asked about any side effects you are experiencing, any new treatments you are having, and if you have needed any blood products. The phone call should take about 10 minutes.

This is an investigational study. Lenalidomide is FDA approved and commercially available. Lenalidomide is approved for the treatment of patients with transfusion-dependent anemia due to low- or intermediate-1-risk myelodysplastic syndromes associated with the chromosome 5 abnormality with or without other chromosome abnormalities. Lenalidomide is also approved in combination with dexamethasone for the treatment of patients with multiple myeloma that have received at least one prior therapy. Its use in this study is investigational. Darbepoetin alfa is approved by FDA for treatment of low red blood cell in patients with cancer and kidney disease. The use of these drugs together is considered to be investigational. Up to 39 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >/=18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Have low or intermediate-1 IPSS risk category MDS (excluding 5q deletion)
5. red blood cell (RBC) transfusion-dependent anemia defined as no transfusion free interval of >/= 56 consecutive days within the past 112 days.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at study entry.
7. Laboratory test results within these ranges: Serum creatinine </= 1.5 mg/dL ,Total bilirubin </= 1.5 mg/dL ,AST (SGOT) and ALT (SGPT) </= 3 x ULN, ANC >/= 500 /uL, Platelet count >/= 30,000/uL (untransfused)
8. Disease free of prior malignancies for >/=2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast
9. Patients who are on epoetin alfa or darbepoetin prior to enrollment will be allowed to enroll if they have failed such therapy, failure defined as transfusion requiring despite >/= 6 weeks of epoetin alfa at dose of 40,000 units/week and darbepoetin alfa at dose of 150 mcg/ 2 week. No washout period will be necessary. Upon study entry patients receiving epoetin alfa will be switched over to darbepoetin.
10. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of prescribing lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
11. continued from #10 Men must agree to use a latex condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy.

Exclusion Criteria:

1. Clinically significant anemia owing to iron, B12, or folate deficiencies.
2. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
3. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide)
4. Concomitant use of steroids will not be allowed unless used for premedication in preparation for transfusions, treatment of hypersensitivity reaction related to lenalidomide or any underlying medical condition other than MDS (e.g. Chronic Obstructive Pulmonary Disease (COPD)).
5. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
6. Use of any other experimental drug or therapy within 28 days of baseline.
7. Known hypersensitivity to thalidomide.
8. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
9. Any prior use of lenalidomide.
10. Concurrent use of other anti-cancer agents or treatments.
11. Known positive for HIV or infectious hepatitis, type A, B or C.
12. Hypersensitivity to darbepoetin or any component of the formulation (including polysorbate 80 and/or albumin);
13. Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 2/22/2009 to 4/20/2010. All patients were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Study terminated due to low accrual, one patient registered on study.
Period: Overall Study
Arm/Group | Lenalidomide + Darbepoetin Alfa
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide + Darbepoetin Alfa
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Transfusion Independence Response
Description: Response defined as transfusion independence (no red blood cell transfusions) for at least 8 weeks, anytime during the six 28-day cycles of therapy.
Time Frame: Over six 28-day cycles (approximately 168 days)
Population: Analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | Lenalidomide + Darbepoetin Alfa
Number analyzed (Participants) | 1
participants | 0

ADVERSE EVENTS:
Time Frame: 1 year 4 months
Arm/Group | Lenalidomide + Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide + Darbepoetin Alfa (N=1)
Neutropenic fever (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide + Darbepoetin Alfa (N=1)
fatigue (General disorders) | 1 (1)
Bilateral edema (Cardiac disorders) | 1 (1)
Bone Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes